CLINICAL TRIAL: NCT00395200
Title: Autologous Adult Human Mesenchymal Stem Cells: a Neuroprotective Therapy for Multiple Sclerosis
Brief Title: Mesenchymal Stem Cells in Multiple Sclerosis (MSCIMS)
Acronym: MSCIMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Peter Connick, Research Associate, University of Cambridge
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRCRG44871; REC Reference: 07/Q0108/104
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Safety; Therapeutics; Mesenchymal Stem Cells; Multipotent Mesenchymal Stromal Cells; Optic Neuritis
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC Treatment (Experimental)
  Interventions: Procedure: MSC Treatment

INTERVENTIONS:
Procedure: MSC Treatment — Intravenous administration of up to 2x10^6 autologous MSCs per kg
  Other Names: Mesenchymal Stem Cells; Multipotent Mesenchymal Stem Cells; Multipotent Mesenchymal Stromal Cells

SUMMARY:
Hypothesis: Intravenous administration of bone marrow-derived autologous adult human mesenchymal stem cells is a safe novel therapeutic approach for patients with multiple sclerosis.

Mesenchymal Stem Cells in Multiple Sclerosis (MSCIMS) is a phase I/IIA trial designed to establish the safety of intravenous administration of bone marrow-derived autologous adult human mesenchymal stem cells to patients with multiple sclerosis.

DETAILED DESCRIPTION:
Disease under investigation: Multiple Sclerosis

Phase: I/IIA

Number of patients: 10

Design: 18 month cross over, single treatment at 6 months

Intervention: Administration of bone marrow-derived autologous mesenchymal stem cells

Route of administration: Intravenous

Dose: Up to 2,000,000 Mesenchymal Stem Cells per kilogram

Source of patients: Referrals accepted from Neurologists in East Anglia and North London, UK

Referral Criteria: (all 3 required)

1. Clinically definite multiple sclerosis
2. Expanded Kurtzke Disability Status Score 2.0 - 6.5 (inclusive)
3. Evidence of optic nerve damage by

   * history of optic neuritis, or
   * relative afferent pupillary defect, or
   * optic atrophy on fundoscopy, or
   * abnormal visual evoked potential from either or both eyes suggestive of demyelination

Primary Objective: Establish the safety of intravenously administered bone marrow-derived autologous mesenchymal stem cells at a dose of up to 2,000,000 cells/kg over 12 months by monitoring adverse reactions.

Secondary Objectives: Explore the efficacy of intravenously administered bone marrow-derived autologous mesenchymal stem cells at a dose of up to 2,000,000 cells/kg over 12 months on visual function by clinical, neurophysiological, and imaging assessments.

Outcome Measures:

1. Primary

   * Adverse events
2. Secondary

   * Visual function (acuity and colour)
   * Visual evoked potential latency
   * Optic nerve Magnetisation Transfer Ratio
   * Retinal nerve fibre layer thickness (by optical coherence tomography)
   * Brain lesion Magnetisation Transfer Ratio
   * MRI brain T1 hypointensity load
   * T cell response suppression
3. Tertiary

   * Multiple Sclerosis Functional Composite Score
   * Expanded Kurtzke Disability Status Score

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite multiple sclerosis
* Expanded Kurtzke Disability Status Score 2.0 - 6.5 (inclusive)
* Evidence of optic nerve damage by:
* history of optic neuritis, or
* relative afferent pupillary defect, or
* optic atrophy on fundoscopy, or
* abnormal visual evoked potential from either or both eyes suggestive of demyelination
* Prolonged visual evoked potential P100 latency with preserved waveform
* T2 lesion on MRI optic nerve
* Retinal nerve fibre layer thickness on optical coherence tomography > 40 microns

Exclusion Criteria:

* Age < 18 years
* Age > 65 years
* Patient lacks capacity to give informed consent
* Presence of a severe bleeding disorder
* Planning a pregnancy during the trial period
* Current MS disease modifying therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | 0,1,2,3,4,12 and 52 weeks post treatment

SECONDARY OUTCOMES:
Visual function (acuity and colour) | 12 and 52 weeks post treatment
Visual evoked potential latency | 12 and 52 weeks post treatment
Optic nerve Magnetisation Transfer Ratio | 12 and 52 weeks post treatment
Retinal nerve fibre layer thickness (by optical coherence tomography) | 12 and 52 weeks post treatment
Brain lesion Magnetisation Transfer Ratio | 12 and 52 weeks post treatment
MRI brain T1 hypointensity load | 12 and 52 weeks post treatment
Multiple Sclerosis Functional Composite Score | 12 and 52 weeks post treatment
Expanded Kurtzke Disability Status Score | 12 and 52 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Siddharthan Chandran, MBChB, PhD, Principal Investigator — University of Cambridge
Locations (2):
- United Kingdom (2):
  - University of Cambridge Dept of Clinical Neurosciences, Cambridge, Cambridgeshire
  - University College London Institute of Neurology, London, London

REFERENCES:
- [Background] Connick P, Kolappan M, Patani R, Scott MA, Crawley C, He XL, Richardson K, Barber K, Webber DJ, Wheeler-Kingshott CA, Tozer DJ, Samson RS, Thomas DL, Du MQ, Luan SL, Michell AW, Altmann DR, Thompson AJ, Miller DH, Compston A, Chandran S. The mesenchymal stem cells in multiple sclerosis (MSCIMS) trial protocol and baseline cohort characteristics: an open-label pre-test: post-test study with blinded outcome assessments. Trials. 2011 Mar 2;12:62. doi: 10.1186/1745-6215-12-62. PMID 21366911
- [Derived] Connick P, Kolappan M, Crawley C, Webber DJ, Patani R, Michell AW, Du MQ, Luan SL, Altmann DR, Thompson AJ, Compston A, Scott MA, Miller DH, Chandran S. Autologous mesenchymal stem cells for the treatment of secondary progressive multiple sclerosis: an open-label phase 2a proof-of-concept study. Lancet Neurol. 2012 Feb;11(2):150-6. doi: 10.1016/S1474-4422(11)70305-2. Epub 2012 Jan 10. PMID 22236384
- See also: University of Cambridge Dept. of Clinical Neurosciences — http://www-neurosciences.medschl.cam.ac.uk
- See also: UCL Institute of Neurology — http://www.ion.ucl.ac.uk
- See also: Study protocol and baseline characteristics of the cohort — http://www.trialsjournal.com/content/12/1/62/abstract